CLINICAL TRIAL: NCT06396715
Title: Optimal Therapeutic Dose of Transcranial Direct Current Stimulation for Functional Upper Limb Recovery in People With Stroke: Multicenter Randomized Clinical Trial
Brief Title: Optimal Therapeutic Dose of tDCS for Functional Upper Limb Recovery in People With Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Maricel Garrido Montenegro, Clinical Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OAIC: 1390/23
Record Dates: First submitted 2024-04-26; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Neurologic Deficits
Keywords: Stroke; Transcranial direct current stimulation; Upper limb; Occupational Therapy
MeSH Terms: conditions — Stroke; Neurologic Manifestations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This methodological design is carried out following the guidelines of the CONSORT 2010 guidelines for clinical trials.
  Study type and design: a two-arm, multicenter, double-blind randomized clinical trial (RCT) is proposed.
  Population: adults with a diagnosis of subacute unihemispheric stroke with motor and functional deficit of the upper limb who attend the Hospital Clínico de la Universidad de Chile (HCUCH) and the Hospital San José (HSJ).
Who Masked: Participant, Care Provider
Masking Description: Patients will be assigned to the 30-minute tDCS with mCIMT or 20-minute tDCS with mCIMT group using block randomization. When the informed consent is signed by the patient, the recruiter will notify the person in charge of randomization (the one who has no relationship with the patient or their medical data) to assign the patient to one of the two groups (called group 1) or group 2), without knowing which corresponds to 30 or 20 minutes of stimulation. Once the group is known, the therapy coordinator will be informed, and make a note of the assigned group (1 or 2) on the patient's record sheet. The patient, the therapists and the evaluators will be kept blinded since they will not know the duration of the stimulation of group 1 or 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-minute tDCS with mCIMT (Experimental): tDCS: the tDCS montage will be of a bi-hemispheric and the stimulation will be applied simultaneously to the upper extremity motor training session carried out in the hospital. There will be a total of 18 sessions with 30 minutes of tDCS stimulation (2 mA intensity), with a frequency of three times a week for six weeks.
  mCIMT: during a period of five days a week, for six weeks, both groups will perform a mCIMT protocol. On days when the patient does not go to the hospital for treatment, they must perform the activities at home with the support of a family member or caregiver if necessary.
  1. Restriction of movements of the unaffected hand through the use of a glove for 6 hours per day: the glove limits the mobility of the fingers but allows free movement of the wrist, elbow and shoulder.
  2. Intensive and individualized training of the affected arm for 2 hours a day.
  Interventions: Device: Transcranial direct current stimulation
- 20-minute tDCS with mCIMT (Active Comparator): tDCS: the tDCS montage will be of a bi-hemispheric and the stimulation will be applied simultaneously to the upper extremity motor training session carried out in the hospital. There will be a total of 18 sessions with 20 minutes of tDCS stimulation (2 mA intensity), with a frequency of three times a week for six weeks.
  mCIMT: during a period of five days a week, for six weeks, both groups will perform a mCIMT protocol. On days when the patient does not go to the hospital for treatment, they must perform the activities at home with the support of a family member or caregiver if necessary.
  1. Restriction of movements of the unaffected hand through the use of a glove for 6 hours per day: the glove limits the mobility of the fingers but allows free movement of the wrist, elbow and shoulder.
  2. Intensive and individualized training of the affected arm for 2 hours a day.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS is a type of non-invasive brain stimulation that in a standard paradigm, low intensity current (1-2 mA) is applied continuously through a battery connected to two 20 to 35 cm2 surface electrodes located on the scalp: an anode and a cathode. In the interhemispheric competition model, tDCS can serve as a means to increase ipsilesional cortical excitability through anodal stimulation, to decrease contralesional cortical excitability through cathodal stimulation, or to do both through a montage of bi-hemispheric electrodes.

SUMMARY:
Stroke is one of the main causes of disability worldwide. The main disability after a stroke is hemiparesis of an Upper Limb (UL), with a prevalence of 70%. Although conventional UL therapies achieve good recovery, their effectiveness is still limited since only 5 to 20% of patients manage to completely recover. This has led to the use of therapies in a combined manner in order to achieve greater benefit. Due to its effects on brain neuroplasticity processes, transcranial direct current stimulation (tDCS), a type of non-invasive brain stimulation, has begun to be used as a complement to standard UL therapies, including combined with Constraint Induced Movement Therapy, whether original or modified (CIMT-mCIMT), with which it shares neurological principles, with evidence of its benefits.

In patients with mild and moderate stroke, tDCS has been used with the aim of reestablishing the altered brain balance by reducing the hyperactivity of the unaffected hemisphere and/or activating the affected hemisphere. A recent meta-analysis mentions that tDCS plus other therapies improve the function of the UL. However, the high heterogeneity of the protocols does not allow us to know the optimal dose, which, in turn, makes decision making in clinical practice difficult. This makes it apropos to develop studies that define therapeutic doses. This would contribute to clinical guidelines and allow to optimize public resources in rehabilitation.

The present study aims to compare the evolution of functional recovery of the UL in people with subacute stroke who attend the Hospital Clínico de la Universidad de Chile and the Hospital San José, after receiving bi-hemispheric tDCS, administered through a protocol of 18 thirty-minute sessions (experimental group) versus a protocol of 18 twenty-minute sessions (active comparator group). The hypothesis is that the experimental group obtains at least 5% more functional recovery compared to the active comparator group. One of the secondary objectives is to identify in which session the recovery plateau is achieved. A randomized, double-blind clinical trial is proposed, where patients will be assigned either to the experimental or active comparator group and both will receive mCIMT as standard therapy. Clinical and socio-demographic information will be gathered and patients will be evaluated with UL motor and functional recovery scales, as well as an evaluation of independence in basic Activities of Daily Living (ADL), among others.

DETAILED DESCRIPTION:
Motor deficit and disability of the upper extremity (US) continues to be the most common sequelae in these patients, which has a significant impact on daily activities. It reduces independence and the probability of returning to work, among others. Although there is a high number of treatments with evidence, patients continue to have sequelae deficits. In addition to this, the high heterogeneity of the protocols makes it difficult to select the best alternative. Therefore, when deciding to use a treatment one of the biggest questions is to determine which combination of therapies and which dose is the most effective.

In the clinical trial carried out by our research team and published in 2022, it was demonstrated that the combination of rehabilitation strategies such as modified Constraint Induced Movement Therapy (mCIMT) and Transcranial Direct Current Stimulation (tDCS), generate significant results in motor and functional recovery of Ul in patients with acute and subacute stroke who are hospitalized. However, there is still no clarity in the optimal (effective and efficient) protocol and dose for subacute patients undergoing outpatient therapy. This is why our proposal aims to answer the pending questions through a randomized clinical trial that includes patients in the subacute stage who have been discharged from the hospital. Furthermore, the optimal dose (stimulation time and number of sessions) would be defined which would allow clear, updated, and accurate evidence to be generated in these patients.

ASSUMPTIONS

* The literature suggests that the best results of UL recovery, in protocols that include tDCS, are obtained with a moderate amount of total number of sessions (comprising between 15-24 sessions), but our local RCT showed results in 7 sessions.
* A very long therapy schedule is uncomfortable for the patient and caregiver and not very feasible to apply in our public health system, which is why the investigators propose an intermediate duration of 18 sessions.

It is reasonable to think that functional recovery tends to stabilize over time and that in a duration of 18 sessions could demonstrate the plateau.

HYPOTHESIS People with subacute stroke and moderate motor deficit of the upper limb who attend outpatient therapy and receive 18 sessions of 30 minutes of Bi-hemispheric Transcranial Direct Current Stimulation obtain at least 5% more functional recovery of the upper limb compared to those people who receive 18 sessions of 20 minutes of stimulation.

GENERAL OBJECTIVE Compare the evolution of functional recovery of the upper limb in people with subacute stroke who attend the Clinical Hospital of the University of Chile and the San José Hospital, after receiving bi-hemispheric transcranial stimulation by direct current, administered through a protocol of 18 30-minute sessions versus a protocol of 18 20-minute sessions.

METHODOLOGY AND PROCEDURES This methodological design is carried out following the guidelines of the CONSORT 2010 guidelines for clinical trials.

Study type and design: a two-arm, multicenter, double-blind randomized clinical trial (RCT) is proposed.

Population: adults with a diagnosis of subacute unihemispheric stroke with motor and functional deficit of the upper limb who attend the Hospital Clínico de la Universidad de Chile (HCUCH) and the Hospital San José (HSJ).

Interventions. Patients will be randomized to one of the following treatment groups: Experimental Group (30 minutes of bi-hemispheric tDCS combined with mCIMT for 18 sessions) or Active comparator Group (20 minutes of bi-hemispheric tDCS combined with mCIMT for 18 sessions).

General procedures.

* During the protocol, patients can continue participating in the usual interdisciplinary rehabilitation program in their hospitals, but it is suggested that they do not add therapies associated with the upper limb while participating in the protocol, as this may generate a risk of injury due to overuse.
* All patients will undergo neuromuscular taping on the deltoid of the paretic shoulder, with weekly changes, since it is part of the usual care at HCUCH.
* Patients should attend therapy wearing comfortable clothing (t-shirt and sweatshirt/shorts).
* Patients should be informed that, if they experience pain or discomfort while performing activities at home, practice should be temporarily suspended and the therapist notified. A transfer package is prepared, which will allow to monitor compliance with the CIMT protocol at home. Some activities of the transfer package include the delivery of videos with therapeutic material and the activities to be performed at home, as well as telephone follow-up to verify compliance with the completion of a check list-type guideline.

ELIGIBILITY:
Inclusion Criteria:

* Single event of ischemic or hemorrhagic unihemispheric stroke, cortical or subcortical.
* Brachial hemiparesis.
* Stroke evolution time greater than 7 days and equal to or less than 90 days.
* Subjects attend rehabilitation at the Hospital Clínico de la Universidad de Chile and Hospital San José.
* Age equal to or greater than 18 years.
* Present some level of UL motor activity: at least 20º of active wrist extension and 10º of finger extension.
* Have a caregiver and/or support network if necessary to attend outpatient therapies, as well as to supervise activities at home.
* Signing of informed consent by the patient.

Exclusion Criteria:

* Prior central stroke with motor sequelae.
* Present severe aphasia with a score ≥ 2 on the language item on the National Institutes of Health Stroke Scale evaluation.
* Severe cognitive impairment, with a score ≤ 15 points on the Mini-mental state examination.
* Present shoulder subluxation and/or pain > 4 points on the visual numerical pain scale.
* History of epilepsy and/or use of antiepileptic drugs.
* Metal implants or pacemakers.
* Pregnancy.
* Any condition that, in the opinion of the doctor, impedes the correct performance of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Functional recovery of upper extremity | 18 days, 3 and 6 months later
  Considers the use of the upper extremity in functional activities and will be evaluated with the Wolf Motor Function Test. Minimum score=0, maximum score=75, higher scores indicating better performance.

SECONDARY OUTCOMES:
Motor recovery of upper extremity | 18 days, 3 and 6 months later
  Considers global sensorimotor functioning of the upper extremity and will be evaluated with Fugl Meyer Assessment Upper Extremity. Minimum score=0, maximum score=66, higher scores indicating better performance.
Independence in activities of daily living | 18 days, 3 and 6 months later
  Considers improvement in functional independence and will be evaluated with Functional Independence Measure. Minimum score=18, maximum score=126, higher scores indicating better performance.
Quality and quantity of movement of the upper limb | 18 days, 3 and 6 months later
  Considers improvement in quality of movement and quantity of use and will be evaluated with Motor Activity Log. Minimum score=0, maximum score=5, higher scores indicating better performance.
Health related quality of life | 18 days, 3 and 6 months later
  Considers effect on quality of life and will be evaluated with Stroke Impact Scale. Minimum score=0, maximum score=100 for domains, higher scores indicating better performance.
Satisfaction with intervention | At the end of the treatment
  Questionnaire that allows you to know the degree of satisfaction with the intervention received. 15 questions, each one has the option to answer: strongly agree, agree, disagree, strongly disagree or neither agree nor disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Maricel Garrido, Principal Investigator — University of Chile

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be available in English and Spanish.
Supporting Information: Study Protocol
Time Frame: For a year.
Access Criteria: Send email to main researcher.

REFERENCES:
- [Result] Pollock A, Farmer SE, Brady MC, Langhorne P, Mead GE, Mehrholz J, van Wijck F. Interventions for improving upper limb function after stroke. Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD010820. doi: 10.1002/14651858.CD010820.pub2. PMID 25387001
- [Result] Garrido M M, Alvarez E E, Acevedo P F, Moyano V A, Castillo N N, Cavada Ch G. Early transcranial direct current stimulation with modified constraint-induced movement therapy for motor and functional upper limb recovery in hospitalized patients with stroke: A randomized, multicentre, double-blind, clinical trial. Brain Stimul. 2023 Jan-Feb;16(1):40-47. doi: 10.1016/j.brs.2022.12.008. Epub 2022 Dec 28. PMID 36584748
- [Result] Jiang L, Xu H, Yu C. Brain connectivity plasticity in the motor network after ischemic stroke. Neural Plast. 2013;2013:924192. doi: 10.1155/2013/924192. Epub 2013 Apr 24. PMID 23738150
- [Result] Grefkes C, Nowak DA, Eickhoff SB, Dafotakis M, Kust J, Karbe H, Fink GR. Cortical connectivity after subcortical stroke assessed with functional magnetic resonance imaging. Ann Neurol. 2008 Feb;63(2):236-46. doi: 10.1002/ana.21228. PMID 17896791
- [Result] Sankarasubramanian V, Machado AG, Conforto AB, Potter-Baker KA, Cunningham DA, Varnerin NM, Wang X, Sakaie K, Plow EB. Inhibition versus facilitation of contralesional motor cortices in stroke: Deriving a model to tailor brain stimulation. Clin Neurophysiol. 2017 Jun;128(6):892-902. doi: 10.1016/j.clinph.2017.03.030. Epub 2017 Mar 21. PMID 28402865
- [Result] Etoom M, Hawamdeh M, Hawamdeh Z, Alwardat M, Giordani L, Bacciu S, Scarpini C, Foti C. Constraint-induced movement therapy as a rehabilitation intervention for upper extremity in stroke patients: systematic review and meta-analysis. Int J Rehabil Res. 2016 Sep;39(3):197-210. doi: 10.1097/MRR.0000000000000169. PMID 27123790
- [Result] Liew SL, Santarnecchi E, Buch ER, Cohen LG. Non-invasive brain stimulation in neurorehabilitation: local and distant effects for motor recovery. Front Hum Neurosci. 2014 Jun 27;8:378. doi: 10.3389/fnhum.2014.00378. eCollection 2014. PMID 25018714
- [Result] Gomez Palacio Schjetnan A, Faraji J, Metz GA, Tatsuno M, Luczak A. Transcranial direct current stimulation in stroke rehabilitation: a review of recent advancements. Stroke Res Treat. 2013;2013:170256. doi: 10.1155/2013/170256. Epub 2013 Feb 27. PMID 23533955